CLINICAL TRIAL: NCT06234566
Title: The Effect of Low Speed Drilling Without Irrigation Versus Conventional Drilling With Irrigation in Extra Short Implants on Primary Stability and Marginal Bone Loss
Brief Title: Effect of Different Drilling Techniques on Primary Stability and Marginal Bone Loss of Extra Short Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Collaborators: Mode Medical Implant Manufacturer (Unknown)
Responsible Party: Principal Investigator, Ömer Faruk Okumuş, Assistant Professor, Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDF-OKUMUS-001
Record Dates: First submitted 2024-01-18; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Different Surgical Techniques in Dental Implant Surgery
Keywords: Dental Implants; Low speed drill; Extra Short Implants; Primary Stability; Marginal Bone Loss; Osstel; Osseointegration
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Speed Drilling Without Irrigation (Experimental)
  Interventions: Procedure: Low Speed Drilling Without Irrigation
- Conventional Drilling with Irrigation (Active Comparator)
  Interventions: Procedure: Conventional dental implant surgery

INTERVENTIONS:
Procedure: Conventional dental implant surgery — It is performed to reconstruct lost teeth. These are surgical procedures performed to place dental implants in the jaw bones. To prepare the implant socket, drilling is performed with serum irrigation at a speed of 800 rpm.
  Arms: Conventional Drilling with Irrigation
Procedure: Low Speed Drilling Without Irrigation — It is performed to reconstruct lost teeth. These are surgical procedures performed to place dental implants in the jaw bones. To prepare the implant socket, drilling is performed at a speed of 50 rpm without serum irrigation.
  Arms: Low Speed Drilling Without Irrigation

SUMMARY:
Our aim in this study is to compare the effects of low-speed drilling surgery technique without irrigation and conventional implant surgery technique with irrigation on extra short implants. The criteria to be taken into consideration when investigating the effect of these techniques on implants are as follows: evaluation of osseointegration at the end of three months, evaluation of marginal bone loss at the end of three months, initial insertion torque values (maximum insertion torque and final insertion torque), ISQ values obtained with a radiofrequency analyzer (Osstel) at the beginning and at the end of three months.

ELIGIBILITY:
Inclusion Criteria:

* There must be toothless space in the maxillary and mandibular posterior region (distal part of the canine in each quadrant).
* The edentulous space should not require additional bone grafting.
* Bleeding areas on probing should be less than 10%
* There should be no pathological periodontal pockets
* Patients who do not smoke or smoke less than 10 cigarettes
* There should be no bruxism
* At least 6 months must have passed since the last tooth extracted from the toothless space where the implant is planned.
* There should be no diabetes.

Exclusion Criteria:

* Having psychological problems
* Smoking more than 10 cigarettes
* Alcohol and drug use
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the status of osseointegration | Three months after the implant is placed in the bone. At the end of three months
  Fusion of the dental implant with the bone at the microscopic level. Osseointegration will be evaluated as successful or unsuccessful. Successful osseointegration is defined by no mobility in the implant, no radiolucency around the implant on radiography, and no pain in the implant. Otherwise, the osseointegration of the implant is considered unsuccessful.
Marginal bone lose | Three months after the implant is placed in the bone. At the end of three months
  It defines the change in the marginal bone level in the neck area of the implant. It is determined by radiographic examination. The initial radiograph is compared with the radiograph at the end of three months. In measurements where the implant platform is the reference point, bone level changes are calculated in mm.

SECONDARY OUTCOMES:
Insertion Torque value | Surgical stage where the implant is placed
  It is the amount of compression of the implant when screwed into the bone. The value detected by the electronic device that screws the implant into the bone cavity during screwing. It is expressed in Newtons.
Implant Stability Quotient (ISQ Value) | 1- Surgical stage where the implant is placed; 2- Three months after the implant is placed in the bone. At the end of three months
  The value obtained by the resonance frequency analysis (RFA) device used to measure the primary stability of dental implants. The RFA technique is based on continual excitation of the implant through dynamic vibration analysis. A transducer is connected to an implant, which is excited over a range of sound frequencies with subsequent measurement of the vibratory oscillation of the implant. It is a non-invasive technique.